CLINICAL TRIAL: NCT06134999
Title: Study of Patients With Knee Prostheses Treated With Noninvasive Neuromodulation. PRONES Trial
Brief Title: Study of Patients With Knee Prostheses Treated With Noninvasive Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRONES
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Knee Prosthesis
Keywords: Total Knee Replacement; physical therapy modality; Electric Stimulation, Transcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Non-invasive Neuromodulation Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7.
  Interventions: Device: Placebo Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 10 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7.
  Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 millivolt and intensity 0.5 μA.
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but microcurrents device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents.
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
It will consist of a randomized clinical trial with a control group. The sample will be distributed as homogeneously as possible into two groups, which will be randomly divided into a control group, to which the usual general treatment will be applied, and an experimental group, which will be treated with the NESA XSignal device. During the procedure, the subjects will continue to receive the usual care routine.

DETAILED DESCRIPTION:
The main objective will be to evaluate the efficacy of the NESA XSignal device in relation to the improvement of pain, functionality and quality of life in patients who have undergone total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Total knee replacement surgery at the Hospital San Juan de Dios de Tenerife.
* Be able to freely consent to take part in the study.

Exclusion Criteria:

* No contraindications for treatment with NXSignal: pacemakers, internal bleeding, poor skin condition with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and/or electricity phobia.
* Patients with total knee prosthesis of more than 3 months of evolution.
* Patients with total knee prosthesis with complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain assessed by VAS | Baseline and up to four weeks
  The instrument will be used to measure the change of pain before and after the intervention will be the Visual Analogue Scale (VAS).
  Participants will be asked to mark the level of their pain on a 100 mm, no hatched VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable".
Change in WOMAC questionnaire | Baseline and up to four weeks
  The WOMAC ( Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire measures quality of life, in terms of Symptomatology and Physical Disability, in people with osteoarthrosis of the hip or knee.
  It contains 24 items grouped into 3 scales: pain (0-20), stiffness (0-8), functional capacity (0-68).
  The scales are used separately, they are not added together.
  Each item is answered with a 5-level verbal-type scale that is coded:
  None = 0; Little = 1; Quite a lot = 2; A lot = 3; Very much = 4.
Change in the quality of life test | Baseline and up to four weeks
  The EuroQol questionnaire will be used: a generic instrument for measuring health-related quality of life that can be used both in relatively healthy individuals (general population) and in groups of patients with different pathologies. The individual him/herself assesses his/her state of health, first in levels of severity by dimensions.
  The descriptive system contains five health dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression) and each has three levels of severity (no problems, some problems or moderate problems, and severe problems).
  severity levels are coded 1 if the response option is "no (I have) problems"; 2 if the response option is "some or moderate problems"; and 3 if the response option is "many problems".

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos del Castillo Rodríguez, PhD, Principal Investigator — Hospital San Juan de Dios Tenerife
Locations (1):
- José Carlos del Castillo Rodríguez, Santa Cruz de Tenerife, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilches C, Sulbaran JD, Fernandez JE, Gisbert JM, Bausili JM, Pelfort X. Fast-track recovery technique applied to primary total hip and knee replacement surgery. Analysis of costs and complications. Rev Esp Cir Ortop Traumatol. 2017 Mar-Apr;61(2):111-116. doi: 10.1016/j.recot.2016.10.002. Epub 2017 Jan 8. English, Spanish. PMID 28073671
- [Background] Jansson MM, Harjumaa M, Puhto AP, Pikkarainen M. Patients' satisfaction and experiences during elective primary fast-track total hip and knee arthroplasty journey: A qualitative study. J Clin Nurs. 2020 Feb;29(3-4):567-582. doi: 10.1111/jocn.15121. Epub 2019 Dec 8. PMID 31769559
- [Background] Mistry JB, Elmallah RD, Bhave A, Chughtai M, Cherian JJ, McGinn T, Harwin SF, Mont MA. Rehabilitative Guidelines after Total Knee Arthroplasty: A Review. J Knee Surg. 2016 Apr;29(3):201-17. doi: 10.1055/s-0036-1579670. Epub 2016 Mar 10. PMID 26963074
- [Background] Davila Castrodad IM, Recai TM, Abraham MM, Etcheson JI, Mohamed NS, Edalatpour A, Delanois RE. Rehabilitation protocols following total knee arthroplasty: a review of study designs and outcome measures. Ann Transl Med. 2019 Oct;7(Suppl 7):S255. doi: 10.21037/atm.2019.08.15. PMID 31728379